CLINICAL TRIAL: NCT06924892
Title: Assessment of Music Experiences in Navigating Depression (AMEND)
Brief Title: Assessment of Music Experiences in Navigating Depression
Acronym: AMEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Carnegie Hall Weill Music Institute (Unknown); Cooper Union College (Unknown); Third Street Music Settlement (Unknown)
Responsible Party: Principal Investigator, Joanne Loewy, Professor/Director, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY-22-01609; 1909623-38 (Other Grant/Funding Number: National Endowment for the Arts)
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Depression
Keywords: Depression; Music Assessment; Music Therapy; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Music therapy or no intervention provided for all consented participants
Who Masked: Participant, Care Provider
Masking Description: Participants were provided options for various music study inclusions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music Therapy (Experimental): Music therapy session for 3 months once a week
  Interventions: Behavioral: Music therapy
- Wellness Concerts (Other): Participants attended wellness concerts.
  Interventions: Other: Wellness Concerts

INTERVENTIONS:
Behavioral: Music therapy — Independent music therapy 45-minute sessions provided weekly for 3 months
  Other Names: Music
  Arms: Music Therapy
Other: Wellness Concerts — Wellness Concerts provided at partner sites (Carnegie Hall Weill Music Institute, Cooper Union College, Third Street Music Settlement).
  Arms: Wellness Concerts

SUMMARY:
The study team sought to scientifically investigate strategic subsets of depressed individuals or people prone to or at-risk of depression through music experiences of individual, group, and blended supported contexts. Meetings with the study multi-disciplinary team, included member of the Carnegie Hall Weill Music Institute and University affiliates, where the study team gathered quantitative and qualitative data in individual and group forums, measuring disease process and levels of participation. Through tabulation of participatory options with standardized depression and resilience measurements, the study team studied how live music could alter depressive symptoms over time and/ or change negative influencers of mood, shift quality of life, and lead toward possibly enhanced disease trajectory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 8-70 years with a clinical diagnosis of Major Depressive Disorder (MOD) who met the DSM-5 (2013) criteria for a Major Depressive Episode, and/or who identify themselves, or are identified by family, or referring clinicians as depressed, or are prone to depression
* Depressive episodes and/or showing symptoms of mild to moderate depression intensity
* Self-reported satisfactory bilateral hearing
* English or Spanish language fluency sufficient to complete the interviews and questionnaires

Exclusion Criteria:

* Axis I diagnosis, aside from MOD, considered the primary diagnosis
* Bipolar Disorder Type I or II,
* Axis II diagnosis such as antisocial or borderline.
* Arrhythmia,
* Pacemaker
* Prolapsed vertebral disc, and
* Recent back or neck injuries.

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Connor-Davidson Resilience Scale (CD-RISC) | end of study at 3 months
  The Connor-Davidson Resilience Scale (CD-RISC) measures inherent resiliency. The 10-item instrument has high internal consistency. Each item consists of a 5-point Likert scale (scored from zero to four). Ranging from 0-40 with higher scores reflecting greater perceived resilience.
The Beck Depression Inventory Second Edition (BDI-II) score | end of study at 3 months
  The Beck Depression Inventory Second Edition (BDI-II) is a multiple-choice self-report inventory that assesses severity of depression. The BDI-II contains 21 items on a 4-point scale from 0 (symptom absent) to 3 (severe symptoms). The minimum score is 0 and the maximum score is 63, with a higher score indicating more severe depressive symptoms.
Child Depression Inventory | end of study at 3 months
  The total score range 0 to 54 which is converted to a T-Score, higher score indicates more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Loewy, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Union Square, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose. To achieve aims in the approved proposal. Proposals should be directed to Joanne.Loewy@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third-party website (Link included in the URL field below)
URL: https://www.mountsinai.org/locations/music-therapy